CLINICAL TRIAL: NCT06836310
Title: The Effect of Virtual Reality Applied to a Task-Oriented Movement on the Upper Extremity for Healthy Individuals: Cross Over Study
Brief Title: Effect of Virtual Reality Applied to a Task-Oriented Movement
Acronym: VR-TOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Zarife Pancar, Assoc.Prof., University of Gaziantep
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GAUN-SBF-PANCAR-04
Record Dates: First submitted 2025-02-08; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Virtual Reality Therapy
Keywords: Virtual reality; upper extremity; reaction time; joint position sense; task-oriented

STUDY DESIGN:
Intervention Model Description: This study is a randomized crossover trial designed to evaluate the effect of virtual reality (VR) applied to a task-oriented movement on upper extremity functions, reaction time, and proprioception in healthy individuals.
  Participants were randomly assigned to one of two sequences:
  f-RP First Group: Performed the task-oriented movement in the real environment first, followed by the VR intervention.
  f-VR First Group: Performed the task-oriented movement in the VR environment first, followed by the real-world intervention.
  Each participant experienced both conditions (real and VR) in a different order, allowing a direct comparison of the interventions within the same individual. The crossover design helps control for individual variability by ensuring that each participant serves as their own control. No period effect or carryover effect was observed in the study, confirming the reliability of the crossover model.
  This model was chosen to better understand how VR-based task-oriente
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real Performance First (f-RP) (Experimental): Participants first performed the task-oriented movement in a real environment. On the following day, they completed the same movement using a virtual reality (VR) system (Oculus Quest 2). Joint Position Sense, Reaction Time, and Gross Manual Dexterity were measured before and after each intervention.
  Interventions: Behavioral: Real Performance Task-Oriented Movement
- Virtual Reality First (f-VR) (Experimental): Participants first performed the task-oriented movement using a virtual reality (VR) system (Oculus Quest 2). On the following day, they completed the same movement in a real environment. Joint Position Sense, Reaction Time, and Gross Manual Dexterity were measured before and after each intervention.
  Interventions: Behavioral: Virtual Reality Task-Oriented Movement

INTERVENTIONS:
Behavioral: Real Performance Task-Oriented Movement — Participants performed a task-oriented movement in a real environment by throwing balls into a physical pool for 10 minutes. The movement was designed to engage upper extremity function.
  Arms: Real Performance First (f-RP)
Behavioral: Virtual Reality Task-Oriented Movement — Participants performed a task-oriented movement in a virtual environment using the Oculus Quest 2 VR system for 10 minutes. The task involved throwing virtual balls into a virtual pool with real-time feedback.
  Arms: Virtual Reality First (f-VR)

SUMMARY:
This study aims to investigate the effect of virtual reality (VR) on upper extremity functions, reaction time, and proprioception in healthy individuals. A randomized crossover design was used, where 26 participants performed a task-oriented movement in both real and virtual environments. Each participant completed a single-session intervention using the Oculus Quest 2 VR system. The study measured Joint Position Sense (JPS), Reaction Time (RT), and Gross Manual Dexterity using standard clinical tests before and after the intervention. The results will help understand how VR-based task-oriented movements influence upper extremity function and whether VR can be effectively used in rehabilitation and sports science applications.

DETAILED DESCRIPTION:
This description provides a summary of the key elements of the study protocol, focusing on the design, interventions, and general approach to evaluation. It does not include the full protocol document or detailed assessment procedures, which are available upon request.

This study is a randomized cross-over trial designed to investigate the acute effects of a task-oriented movement-based virtual reality (VR) application on upper extremity functions in healthy individuals. The primary aim is to evaluate the impact of VR-supported movement exercises on joint position sense (JPS), reaction time (RT), and gross manual dexterity.

The research involves 26 healthy participants who were randomly assigned to two intervention sequences:

Real Performance first (f-RP) group: Participants performed task-oriented movements in a real environment on the first day, followed by a VR-based task-oriented movement session on the second day.

Virtual Reality first (f-VR) group: Participants performed VR-based task-oriented movements on the first day, followed by a real environment session on the second day.

Each intervention lasted 10 minutes and included a task-oriented ball-throwing activity, where participants used repetitive wrist and upper limb movements to throw balls into a target pool placed 2 meters away. The VR intervention was delivered using the Oculus Quest 2 head-mounted display, with real-time visual, auditory, and tactile feedback integrated into the application. The real-world intervention matched the VR setup as closely as possible, including chair position, distance to the target, and ball size.

Assessments were conducted immediately before and after each intervention to observe acute effects. The primary focus was on changes in upper extremity functions and neuromuscular responses following task-oriented movements in VR and real environments.

Data were analyzed for within-group and between-group differences, as well as potential carryover and period effects, using parametric statistical methods appropriate for cross-over trials. The results indicated that VR-based task-oriented applications acutely enhanced reaction time and supported hand functions in healthy individuals. JPS measures remained stable across both intervention types, suggesting that VR-created movement perception can closely resemble real-world joint positioning.

These findings contribute to understanding the short-term effects of VR applications on upper extremity functions and support the potential for VR-based interventions in rehabilitation and performance enhancement.

ELIGIBILITY:
Inclusion Criteria:

* to be over 18 years old,
* volunteering to participate in the study,
* having no upper extremity orthopedic disease (carpal tunnel syndrome, etc.).

Exclusion Criteria:

* not having an upper extremity injury in the last year,
* the presence of rheumatic disease,
* pregnancy,
* the presence of cervical disc herniation and thoracic outlet syndrome.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Reaction Time (RT) in milliseconds | Day 1 (immediately after intervention) and Day 2 (immediately after intervention)
  Reaction time was measured using a mobile application ("Reaction Time Test" app) before and after the intervention. Participants tapped the screen as quickly as possible when a visual stimulus appeared. The average reaction time (in milliseconds) over 25 trials was recorded.

SECONDARY OUTCOMES:
Joint Position Sense (JPS) measured in degrees | Day 1 (immediately after intervention) and Day 2 (immediately after intervention)
  Joint position sense was evaluated using a universal goniometer for both shoulder and wrist proprioception. Participants were asked to reproduce specific joint angles without visual feedback, and the absolute angular error (in degrees) was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Faculty of Sport Sciences, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data (reaction time, joint position sense, and Box and Block Test scores) will be shared upon reasonable request. Data will be available after study completion for researchers conducting related studies. Requests should be submitted via email to z_pancar@hotmail.com
Supporting Information: Study Protocol, SAP
Time Frame: Start Date: Data will be available after study completion. End Date: Data will be available for 5 years after study completion.
Access Criteria: De-identified participant data will be available to researchers conducting related studies in the fields of virtual reality, motor control, proprioception, and reaction time.
  The shared data will include:
  Reaction time (RT) measurements Joint position sense (JPS) measurements Box and Block Test (BBT) scores How can they access it?
  Researchers must submit a formal request explaining their research purpose and how they plan to use the data.
  Requests should be sent via email to [z_pancar@hotmail.com]. URL will be available upon data publication on OSF. Approved researchers will receive access to the de-identified dataset via the Open Science Framework (OSF) repository.
  A direct link to the dataset will be provided upon approval.
URL: https://osf.io/